CLINICAL TRIAL: NCT01556165
Title: Randomised, Double-blind, Parallel-group, Placebo-controlled, Fixed-dose Study of Rasagiline in Early Parkinson's Disease Patients Not Treated With Levodopa in China
Brief Title: Rasagiline in Early Parkinson's Disease Patients Not Treated With Levodopa in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13485A
Record Dates: First submitted 2012-03-13; First posted 2012-03-16 (Estimated); Results first posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Parkinson's Disease
Keywords: Rasagiline; Azilect; Parkinson´s Disease; Motor fluctuations
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rasagiline (Experimental)
  Interventions: Drug: rasagiline
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rasagiline — 1 mg/day, tablets, once daily, orally
  Other Names: Azilect
  Arms: rasagiline
Drug: placebo — tablets, once daily, orally
  Arms: placebo

SUMMARY:
Rasagiline has been developed for the treatment of Parkinson's Disease (PD), as monotherapy in early PD patients not treated with levodopa, and as adjunct therapy to levodopa in levodopa-treated PD patients with motor fluctuations.

The rationale for conducting this study is to evaluate the efficacy, tolerability, and safety of rasagiline compared to placebo in Chinese PD patients not treated with levodopa.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic PD.
* Patients with a Modified Hoehn and Yahr stage <3.

Exclusion Criteria:

* Patients with a clinically significant or unstable medical or surgical condition that would preclude his/her safe and complete study participation.
* Patients with a clinically significant or unstable vascular disease.
* Patients with a clinically significant psychiatric illness, including a major depression, which compromises their ability to provide consent or participate fully in the study.
* Patients with a Mini Mental State Examination (MMSE) score ≤24.
* Patients with a diagnosis of melanoma or a history of melanoma, or a suspicious lesion.

Other inclusion and exclusion criteria may apply.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Principal Investigator — LundbeckClinicalTrials@lundbeck.com
Locations (15):
- China (15):
  - CN015, Beijing
  - CN001, Beijing
  - CN011, Chengdu
  - CN003, Guangzhou
  - CN005, Guangzhou
  - CN017, Guangzhou
  - CN004, Hangzhou
  - CN012, Shanghai
  - CN007, Shanghai
  - CN013, Shanghai
  - CN006, Suzhou
  - CN009, Wuhan
  - CN016, Wuhan
  - CN010, Xi'an
  - CN014, Xi'an

REFERENCES:
- [Derived] Zhang Z, Wang J, Chen S, Liu C, Zhang B, Peng R, Sun S, Sun X, Zhao G, Qu Q, Li Y, Zhu S, Pan X, Shao M, Wang Y. Efficacy and safety of rasagiline in Chinese patients with early Parkinson's disease: a randomized, double-blind, parallel, placebo-controlled, fixed-dose study. Transl Neurodegener. 2018 Dec 6;7:32. doi: 10.1186/s40035-018-0137-5. eCollection 2018. PMID 30534374

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatients aged 35 years or older, who had idiopathic Parkinson's disease and were not treated with levodopa or other antiparkinsonian medications, were recruited for this study from China.
Pre-assignment Details: A Screening Visit was held approximately 28 days prior to group assignment (group assignment was held during the Baseline Visit). Patients who met each of the inclusion criteria and none of the exclusion criteria were eligible to participate in this study.
Period: Overall Study
Arm/Group | Placebo | Rasagiline
Started | 65 | 65
Completed | 53 | 58
Not Completed | 12 | 7
Not completed — Adverse Event | 5 | 3
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal of Consent | 7 | 1

BASELINE CHARACTERISTICS:
Population: The all-patients-treated set (APTS) comprises all randomised patients who took at least one dose of IMP.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rasagiline | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (9.22) | 58.5 (8.72) | 59.0 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 30 | 55
  Male | 40 | 35 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 65 | 65 | 130
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 26 in UPDRS Total Score
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) is a 42-item rating scale designed to assess Parkinson's disease-related disability and impairment. The scale comprises four parts: Part I evaluates mentation, behaviour, and mood symptoms; Part II evaluates activities of daily living (ADL); Part III evaluates motor function; and Part IV evaluates complications of dopaminergic therapy. The total score is the sum of the subscale scores for Parts I to III and ranges from 0 (no disability) to 176 (total dependence).
Time Frame: Baseline to Week 26
Population: The full-analysis set (FAS) comprised all patients in the APTS who had a valid baseline assessment and at least one valid post-baseline assessment of the primary efficacy variable.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Rasagiline
Number analyzed (Participants) | 63 | 64
units on a scale | -0.18 (0.98) | -3.18 (0.95)
Statistical Analysis 1: Comparison: Placebo vs Rasagiline; This study was designed to show a trend, that is, to show a clinical difference in the primary efficacy analysis, at a two-sided significance level of 0.25. Assuming a difference between rasagiline and placebo of a 3-point change in the UPDRS total score and a standard deviation on the change from baseline of 7 points, a sample size of 60 patients per treatment group gave an 88% probability of showing a trend. LOCF (last observation carried forward) was used; Test type: Superiority or Other; p = 0.0254, ANCOVA — No adjustments for multiple comparisons were made; Mean Difference (Final Values) = -3.00, 75% CI 2-sided [-4.53 to -1.47], Standard Error of Mean 1.32

2. Secondary Outcome: Change From Baseline to Week 26 in Subscale Scores of the UPDRS (Part I)
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) Part I evaluates mentation, behaviour and mood symptoms, it comprises 4 parts and the score ranges from 0 (normal) to 16 (severe impairement)
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Rasagiline
Number analyzed (Participants) | 63 | 64
units on a scale | 0.08 (0.15) | -0.54 (0.15)
Statistical Analysis 1: Comparison: Placebo vs Rasagiline; LOCF (last observation carried forward) was used; Test type: Superiority or Other; p = 0.0032, ANCOVA; The same ANCOVA methodology as for the primary endpoint was used; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-1.03 to -0.21], Standard Error of Mean 0.21

3. Secondary Outcome: Change From Baseline to Week 26 in Subscale Scores of the UPDRS (Part II)
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) Part II evaluates activities of daily living, it comprises 13 parts and the score ranges from 0 (normal) to 52 (severe impairement and disability)
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Rasagiline
Number analyzed (Participants) | 63 | 64
units on a scale | 0.25 (0.38) | -0.43 (0.37)
Statistical Analysis 1: Comparison: Placebo vs Rasagiline; LOCF (last observation carried forward) was used; Test type: Superiority or Other; p = 0.1963, ANCOVA; The same ANCOVA methodology as for the primary endpoint was used; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-1.70 to 0.35], Standard Error of Mean 0.52

4. Secondary Outcome: Change From Baseline to Week 26 in Subscale Scores of the UPDRS (Part III)
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) Part III evaluates motor function, it comprises 14 parts and the score ranges from 0 (normal) to 108 (severe impairement and disability)
Time Frame: Baseline to Week 26
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Rasagiline
Number analyzed (Participants) | 63 | 64
units on a scale | -0.52 (0.68) | -2.23 (0.65)
Statistical Analysis 1: Comparison: Placebo vs Rasagiline; LOCF (last observation carried forward) was used; Test type: Superiority or Other; p = 0.0641, ANCOVA; The same ANCOVA methodology as for the primary endpoint was used; Mean Difference (Final Values) = -1.71, 95% CI 2-sided [-3.52 to 0.10], Standard Error of Mean 0.91

5. Secondary Outcome: Time to Onset of Levodopa Therapy
Description: It was stated in the statistical analysis plan (SAP) that if >10% of FAS patients were considered to have taken levodopa during the treatment period, the endpoint, time to onset of levodopa treatment was to be analysed. However, since only one patient (in the placebo group) had levodopa administered during the treatment period, this endpoint was not analysed, as had been defined a priori in the SAP.
Time Frame: Baseline to Week 26
Reporting Status: Not Posted

6. Secondary Outcome: Levodopa Administration Within 26 Weeks
Description: It was stated in the statistical analysis plan (SAP) that if >10% of FAS patients were considered to have taken levodopa during the treatment period, the endpoint, levodopa administration within 26 Weeks was to be analysed. However, since only one patient (in the placebo group) had levodopa administered during the treatment period, this endpoint was not analysed, as had been defined a priori in the SAP.
Time Frame: Baseline to Week 26
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 weeks
Arm/Group | Placebo | Rasagiline
Serious Adverse Events (participants affected / at risk) | 4/65 | 0/65
Other Adverse Events (participants affected / at risk) | 6/65 | 8/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Rasagiline (N=65)
Cataract (Eye disorders) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Rasagiline (N=65)
Accidental overdose (Injury, poisoning and procedural complications) | 3 | 4
Parkinson's disease (Nervous system disorders) | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No